CLINICAL TRIAL: NCT07366892
Title: Fluorescence Visualization and Image Quality Evaluation of Digital Visualization of Suspected Grade III and/or IV Gliomas During Neurosurgery (Leica GLOW400)
Brief Title: Leica Microsystems Sponsored PMCF Study to Collect and Confirm Clinical Data on the Performance of the GLOW400 Device When Used in Accordance With Its Intended Use
Acronym: IMED-GLOW400
Status: Not yet recruiting | Type: Observational
Sponsor: Leica Microsystems (Schweiz) AG (Industry)
Responsible Party: Sponsor
Other Study IDs: GLOW400-PMCFSTUDYPLAN-202501
Record Dates: First submitted 2026-01-07; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Suspected Grade III and IV Gliomas Requiring Surgical Intervention; Neurosurgical Procedure; Glioma; Glioblastoma (GBM)
Keywords: GLOW400; ARveo8x; Digital surgical microscope; 5-ALA fluorescence; Image quality assessment; Grade III gliomas; Grade IV gliomas; High-grade glioma; fluorescence-guided surgery
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GLOW400
  Interventions: Device: GLOW400 is a digital surgical microscope accessory used in fluorescent visualization of suspected grade III or IV gliomas during neurosurgery.

INTERVENTIONS:
Device: GLOW400 is a digital surgical microscope accessory used in fluorescent visualization of suspected grade III or IV gliomas during neurosurgery. — The digital surgical microscope accessory GLOW400 is using the optical excitation and emission filtering of the FL400. The FL400 provides an illumination filter (380nm - 430nm) which when engaged into the light source path of the surgical operating microscope provides, via a light guide, a fluorescence excitation light system used in conjunction with an approved tumor-selective substance (fluorophore) (e.g. Protoporphyrin IX (PpIX) which is resulting of the metabolization of 5-ALA (5 - aminolaevulinic acid)) for tissue characterization in the open neurosurgery field. PpIX is strongly fluorescent with a peak at λ=635 nm as red-violet after excitation with blue light (λ=380-410 nm). The digital surgical microscope accessory GLOW400 is using the optical excitation and emission filtering of the FL400. The fluorescence signal visualized depicts the distribution of the dye in the patient's tissues during the surgical procedure.

SUMMARY:
This post-market clinical follow-up (PMCF) study aims to confirm the safety and performance of the GLOW400 surgical microscope accessory when used in conjunction with the ARveo8x surgical microscope. The study evaluates fluorescence visualization and image quality during standard surgical procedures in neurosurgery. It is a non-interventional, observational study conducted in routine care settings across multiple European sites.

DETAILED DESCRIPTION:
The IMED-GLOW400 study is a prospective, observational, non-interventional clinical investigation conducted in the European Economic Area and Switzerland. It involves the use of the GLOW400 accessory, which digitally enhances fluorescence signals during neurosurgery, providing improved anatomical visualization and contrast. The study compares GLOW400 with the benchmark FL400 optical filter system.

The primary objective is to confirm the image quality and fluorescence visualization performance of GLOW400. Secondary objectives include validating product claims and assessing user experience and safety. An exploratory objective evaluates the extent of tumor resection using volumetric analysis of pre- and post-operative MRI scans.

Data will be collected through structured questionnaires, histopathology confirmation, optional resection forms, and intraoperative video recordings. The study will enroll 37 patients, with at least 29 complete datasets required for analysis. The duration of the study is estimated at 5 to 6 months, with each patient participating only during the surgical procedure.

The study complies with ISO 14155:2020, GDPR, and the Declaration of Helsinki. Ethics Committee approval and informed consent are mandatory prior to enrollment. No additional procedures beyond standard of care are introduced, and risks are limited to those associated with routine surgical practice.

ELIGIBILITY:
Candidates for the for the IMED-GLOW400 Study must be appropriate patients for surgical interventions with suspected intracranial high-grade glioma evidenced by preoperative imaging modalities and have to fulfil all of the following inclusion criteria to be eligible for the recruitment of the study.

Inclusion Criteria

1. Participants must be 18 years of age or older at the time of signing the informed consent.
2. Participants must have suspected high-grade glioma (WHO grade III-IV) as evidenced by preoperative imaging modalities, which require surgical intervention.
3. The active substance 5-aminolevulinic acid (5-ALA) fluorescence dye is administered according to the 5-ALA instructions for use.
4. The participant or their legal representative must understand the study and have voluntarily signed and dated the Informed Consent Form, which has been approved by the Sponsor and the Ethics Committee for this study.

Note for Switzerland only:

Enrollment via legal representative is not permitted. Therefore, only patients who are capable of providing informed consent themselves will be eligible for inclusion in Switzerland.

Exclusion Criteria

1. Known allergy to 5-ALA hydrochloride or protoporphyrin.
2. Patients with porphyria (a condition characterized by the inability to break down protoporphyrin).
3. Any uncontrolled systemic condition that may adversely affect the surgical outcome.
4. Patients holding United States citizenship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population will include patients with suspected grade III or IV gliomas requiring surgical intervention, and who meet the Inclusion/Exclusion Criteria for the IMED-GLOW400 Study.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Flourescence visibility | Periprocedural
  Performance will be evaluated using Questionnaire, a structured Likert-scale survey completed by the operating surgeon during and after surgery.
  The questionnaire assesses:
  1. perceived intensity of fluorescence
  2. perceived volume/ shape and relative location
  3. perceived distribution of fluorescence
  4. anatomical and fluorescence observation (GLOW400 Anatomy only)
  Each item is rated on a 5-point Likert scale:
  1. = Not available
  2. = Insufficient
  3. = Sufficient
  4. = Very good
  5. = Excellent
  Higher scores indicate better performance.
  The outcome is considered acceptable if all ratings are ≥3 (Sufficient or better).
Image quality | Periprocedural
  Performance will be evaluated using Questionnaire, a structured Likert-scale survey completed by the operating surgeon during and after surgery. The questionnaire assesses::
  1. Stereoscopic Perception (3D Depth perception)
  2. Resolution
  3. Noise
  4. Latency
  Each item is rated on a 5-point Likert scale:
  1. = Not available
  2. = Insufficient
  3. = Sufficient
  4. = Very good
  5. = Excellent
  Higher scores indicate better performance.
  The outcome is considered acceptable if all ratings are ≥3 (Sufficient or better).
Anatomy of the brain, including Vessels (GLOW400 Anatomy only) | Periprocedural
  Performance will be evaluated using Questionnaire, a structured Likert-scale survey completed by the operating surgeon during and after surgery. The questionnaire assesses:
  1. Neuroanatomy structures
  2. Vascular structures 4. Perceived contrast (GLOW400 HiFluo only) 5. Bleeding visibility (GLOW400 Anatomy only) 6. Traces of remaining fluorescence (GLOW400 HiFluo only)
  Each item is rated on a 5-point Likert scale:
  1. = Not available
  2. = Insufficient
  3. = Sufficient
  4. = Very good
  5. = Excellent
  Higher scores indicate better performance.
  The outcome is considered acceptable if all ratings are ≥3 (Sufficient or better).

SECONDARY OUTCOMES:
The secondary objectives of this Post-Market Clinical Follow-up (PMCF) study are to assess the continued safety of the device. | Postoperatively
  Safety will be evaluated using Questionnaire B, completed postoperatively by the surgical team. It captures:
  1. Dizziness through using digital 3D visualization
  2. Delayed, interrupted or hindered surgery due to different causes
  3. Occurred injuries to the patient
  4. Breach of sterility
  5. Any patient or user tissue burn event reported.
  6. Confirm user experience with the use of the device in real clinical practice, supporting the marketing claims:
     1. Confidence in decision
     2. Focus during procedure
     3. Surgical course of action
     4. User experience
     5. Mental fatigue
  Responses are binary:
  1. = Yes (event occurred)
  2. = No (event did not occur)
  Lower scores (2 = No) indicate better safety outcomes.
  The outcome is acceptable if no safety events are reported.

OTHER OUTCOMES:
Assessment of the extent of tumor resection | Postoperatively
  The extent of tumor resection will be evaluated using volumetric analysis. The volumetric measurement will be carried out by a neuroradiologist. Precise three-dimensional (3D) rendering and analysis of pre-operative and post-operative MRI images, facilitating accurate assessment of residual tumor volume.
  Radiology reports include:
  • Residual tumor percentage %.
  Based on the residual tumor percentage, the appropriate category will be selected (4):
  * Complete tumor resection: (100% + 0 cm3 CE)
  * Near total resection: (≥ 95% + ≤ 1 cm3 CE)
  * Subtotal resection: (≥ 80% + ≤ 5 cm3 CE)
  * Partial resection: (< 80% ± >5 cm3 CE)

CONTACTS AND LOCATIONS:
Locations (2):
- Unidade Local de Saúde de São João, Porto, Portugal
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication.
Supporting Information: Study Protocol, CSR